CLINICAL TRIAL: NCT07008547
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Profile and Immunogenicity of Subcutaneous Netakimab in Chinese Adult Patients With Moderate to Severe Plaque Psoriasis
Brief Title: To Evaluate the Efficacy and Safety of Netakimab in Chinese Patients With Moderate to Severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SPH-BIOCAD (HK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-085-CN01
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — netakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Netakimab (Experimental): Netakimab administered by subcutaneous injection until Week 52
  Interventions: Biological: Netakimab
- Placebo (Placebo Comparator): Placebo administered by subcutaneous injection until Week 12 then Netakimab subcutaneous injection until 52 week
  Interventions: Biological: Netakimab; Drug: Placebo

INTERVENTIONS:
Biological: Netakimab — Netakimab administered subcutaneously
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to To evaluate the efficacy of subcutaneous (SC) Netakimab in adult Chinese patients with moderate to severe plaque psoriasis. Researchers will compare Netakimab to placebo to see if Netakimab works to treat plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients must voluntarily sign and date an Informed Consent Form (ICF) approved by the Ethics Committee (IEC) prior to any study-related procedures. The legal representative may also be asked to sign the ICF in accordance with local laws and regulations if necessary.

  2) Male or female, ≥ 18 years old at the time of signing the ICF. 3) Patients with plaque psoriasis diagnosed at least for 6 months prior to signing the ICF.

  4) Patients who have inadequate response or intolerance to phototherapy or systemic drug therapy (biological or non-biological agents other than IL-17/IL-17R inhibitors) for psoriasis, or meet the above treatment indications in the opinion of the investigator.

  5) Patients with psoriasis involved body surface area (BSA) of 10% or more, PASI score of 10 or more, and sPGA score of 3 or more at screening.

  6) WOCBP have a negative serum pregnancy test (no pregnancy test is required for women of non-childbearing potential).

  7) Patients of childbearing potential and their partners must implement reliable contraceptive measures as specified in the protocol from signing the ICF until 20 weeks after the last dose of study treatment (see Appendix 10 for details).

  8) Patients who have the ability to follow protocol procedures as judged by the investigator.

Exclusion Criteria:

* 1) Patients with other types of psoriasis (e.g., erythrodermic psoriasis, pustular psoriasis, guttate psoriasis) or any other skin disorders (e.g., eczema) that may affect the treatment/evaluation of psoriasis, and patients with drug-induced psoriasis or a history of drug-induced psoriasis at screening.

  2) Patients who are unable or unwilling to undergo repeated subcutaneous injection and venipuncture (e.g., because of poor tolerability or lack of venous access).

  3) Patients who have received the prohibited drugs or vaccines as specified in the protocol: 4) Patients with hepatitis B virus (HBV) infection, hepatitis C virus (HCV) infection, human immunodeficiency virus (HIV) infection, treponema pallidum (TP) infection.

  5) Patients meeting any of the following criteria for laboratory tests at screening: serum creatinine (Cr) > 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) > 2.5 × ULN; total bilirubin (TBIL) > 1.5 × ULN; white blood cell (WBC) count < 3.0 × 109/L; absolute neutrophil count (ANC) < 2.0 × 109/L; platelet (PLT) count < 100 × 109/L; hemoglobin (Hb) < 90 g/L.

  6) Patients with any psychiatric disorders, including serious depressive disorder, or history of strong suicidal ideation or suicide intention; or clinically significant symptoms of depression (Beck score ≥ 16 at screening), which require intervention treatment determined by a specialist.

  7) Patients with history or evidence of alcohol or drug abuse. 8) Patients with active tuberculosis infection or history of tuberculosis, or current latent tuberculosis infection [positive for interferon gamma release assay (QuantiFERON TB-Gold or T-SPOT etc.)].

  9) Patients with other diseases that may affect the assessment of psoriasis or any other underlying disease (including, but not limited to, clinically significant cardiac, hepatic, renal, respiratory, immune, neurological, endocrine, metabolic, blood, gastrointestinal, or psychiatric disorders) that, in the opinion of the investigator, study treatment may place the patient at additional risks 10) Patients with current or previous malignant tumor within the past 5 years [except adequately treated (cured) squamous cell carcinoma or basalioma, cervical uteri cancer in situ or in situ breast ductal carcinoma].

  11) Patients with known history of serious allergies (allergies to two or more drugs or systemic allergic reactions).

  12) Patients with known allergies or intolerance to monoclonal antibody drugs or any other component of the investigational product or placebo.

  13) Patients who have had major surgery within 30 days prior to screening or scheduled for major surgeries at any time during the study.

  14) Patients with active infection or medical history: 15) Patients with epileptic seizure or the history of epileptic seizure. 16) Patients who are pregnant, breastfeeding, or planning pregnancy at the time of study participation.

  17) Patients who have participated in any other clinical study or within 3 months prior to signing the ICF or are concurrently participating in other clinical studies.

  18) Patients who have other conditions that are not suitable for participation in the study in the judgment of the investigat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving PASI75 | at week 12
  Proportion of subjects with a Psoriatic Area and Severity Index (PASI) score improved by at least 75% (to achieve a PASI 75 response) relative to the baseline PASI score at Week 12
Proportion of subjects achieving sPGA0/1 | at week 12
  Proportion of subjects with a sPGA(Static Physician Global Assessment) either 0 or 1 at Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI75 | through out the study(From baseline to Week 62)
  Proportion of subjects with a Psoriatic Area and Severity Index (PASI) score improved by at least 75% (to achieve a PASI 75 response) relative to the baseline PASI score through out the study
Proportion of subjects achieving PASI90 | through out the study(From baseline to Week 62)
  Proportion of subjects with a Psoriatic Area and Severity Index (PASI) score improved by at least 90% (to achieve a PASI90 response) relative to the baseline PASI score through out the study
Proportion of subjects achieving PASI100 | through out the study(From baseline to Week 62)
  Proportion of subjects with a Psoriatic Area and Severity Index (PASI) score improved by at least100% (to achieve a PASI100 response) relative to the baseline PASI score through out the study
Proportion of subjects achieving PGA | through out the study(From baseline to Week 62)
  Proportion of subjects with a sPGA(Static Physician Global Assessment) either 0 or 1 through out the study
Changes from baseline in NAPSI score | through out the study(From baseline to Week 52)
  Changes from baseline in NAPSI score through out the study

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No